CLINICAL TRIAL: NCT01587066
Title: Efficacy of Quetiapine XR Versus Divalproex on Clinical Outcome Quality of Sleep and Quality of Life in Bipolar Depression
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Bo-Hyun Yoon (Other)
Responsible Party: Sponsor-Investigator, Bo-Hyun Yoon, Doctor, Naju National Hospital
Organization: Naju National Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1443L00059
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine fumarate (Active Comparator)
  Interventions: Drug: Quetiapine fumarate
- Divalproex sodium (Active Comparator)
  Interventions: Drug: Divalproex sodium

INTERVENTIONS:
Drug: Quetiapine fumarate — Efficacy of Quetiapine XR vs. Divalproex on Clinical Outcome, Quality of Sleep and Quality of Life in Bipolar Depression
  Other Names: Seroquel XR, Quetiapine fumarate
  Arms: Quetiapine fumarate
Drug: Divalproex sodium — Efficacy of Quetiapine XR vs. Divalproex on Clinical Outcome, Quality of Sleep and Quality of Life in Bipolar Depression
  Other Names: Depakote XR, Divalproex sodium
  Arms: Divalproex sodium

SUMMARY:
Quetiapine is one of atypical antipsychotics with good efficacy and better side effect profiles than conventional antipsychotics, so it is being widely used beyond the treatment of schizophrenia. Recently, the BOLDER I and II study showed that quetiapine monotherapy is an effective and well-tolerated treatment for depressive episodes in bipolar disorder. However, most c1inicians did not have confidence with quetiapine monotherapy yet, and most practice guidelines recommend the monotherapy with mood stabilizer as the first-line treatment. The Korean medication algorithm for bipolar disorder published in 2006 also recommend the monotherapy with lithium, divalproex, or lamotrigine in the treatment of mild to moderate depressive episode of bipolar disorder.

Therefore, the aim of this study is investigating the efficacy and safety of quetiapine monotherapy when compared with mood stabilizer monotherapy. In addition, the investigators are going to reveal the quality of sleep and quality of life, of the two groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* A diagnosis of Bipolar depression by Diagnostic and Statistical Manual of Mental Disorders- Fourth Edition (DSM-IV)
* Females and males aged 20 to 65 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin (HCG) test at enrollment
* Able to understand and comply with the requirements of the study
* HAM-D score at Visit 0 and Visit 1 should be above 20.
* Willingness to adhere to the schedule of assessments
* Able and willing to comply with self-administration of study drug, or have consistent help or support available

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis 1 disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate or divalproex, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erγthromycin， clarithromycin, troleandomycin, indinavir, nelfinavir，ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin， St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation
* Substance or alcohol dependence at enrollment (except dependence in full remission,and except for caffeine or nicotine dependence) ， as defined by DSM-IV criteria
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 8 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e,g, congestive heart failure,angina pectoris, hypertension) as judged by the investigator Invo1vement in the planning and conduct of the study
* Previous enrollment or randomisation of treatment in the present study.
* Participation in another drug trial within 8 weeks prior enrollment into this study or longer in accordance with local requirements

A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

* Unstable DM defined as enrolment glycosylated hemoglobin (HbAlc) > 8.5%
* Admitted to hospital for treatment of DM or DM related illness in past 12 weeks
* Not under physician care for DM
* Physician responsib1e for patient's DM care has not indicated that patient's DM is controlled
* Physician responsible for patient's DM care has not approved patient's participation in the study
* Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to randomisation. For thiazolidinediones (glitazones) this period should not be less than 8 Weeks
* Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study

  * An absolute neutrophil count (ANC) of s 1.5 x 109 per liter

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
In between the two drugs at baseline MADRS score change at 8 weeks comparison. | one year
  Quetiapine fumarate XR vs. Divalproex sodium treatment compared clinical outcomes in bipolar depression.

SECONDARY OUTCOMES:
Improvement compared with the Number of subjects responding to drug and reliability, and tolerability between the two drugs, quality of sleep and quality of life | one year
  Improvement compared with the Number of subjects responding to drug and reliability, and tolerability between the two drugs, quality of sleep and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Hyun Yoon, Doctor, Principal Investigator — Naju National Hospital
Locations (1):
- Naju National Hospital, Naju, Jeollanam-do, South Korea